CLINICAL TRIAL: NCT05560997
Title: Machine Learning to Identify Metabolic Subtypes of Non-Alcoholic Fatty Liver Disease
Brief Title: Metabolic Subtypes of Non-Alcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yan Bi (Other)
Responsible Party: Sponsor-Investigator, Yan Bi, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Other Study IDs: NAFLDcluster
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2023-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Machine Learning
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- biopsy-proved NAFLD cohort: NAFLD is defined as the presence of at least 5% steatosis based on histological examination.
  Interventions: Diagnostic Test: 10-year ASCVD risk estimation
- longitudinal physical examination cohort: The diagnosis of NAFLD was based on imaging evaluation.
  Interventions: Diagnostic Test: 10-year ASCVD risk estimation

INTERVENTIONS:
Diagnostic Test: 10-year ASCVD risk estimation — High CVD risk was defined as a history of CVD or a 10-year ASCVD risk ≥10%. The 10-year ASCVD risk estimation was carried out according to 2016 Chinese guidelines for the management of dyslipidemia in adults.

SUMMARY:
The purpose of this study was to use machine learning to explore a more precise classification of NAFLD subgroups towards informing individualized therapy.

DETAILED DESCRIPTION:
Clinical characteristics of NAFLD are heterogenous, but current classification for diagnosis is simply based on pathological examination. The conventional pathological classification is insufficient to reflect the complexity and heterogeneity of NAFLD and can not predict the prognosis. Towards precision treatment, a more refined metabolic classification of NAFLD phenotypes is highly demanded for a personalized diagnosis, aiming to identify patients at elevated risk of cardiovascular disease or cirrhosis. This kind of refined classification can provide a more precise diagnosis and enable more individualized preventive interventions and early treatments. In a cross-sectional cohort, unsupervised machine learning was used to cluster patients with biopsy-proved NAFLD from Drum Tower Hospital Affiliated to Nanjing University Medical School based on clinical variables. Verification of the clustering was performed in a longitudinal cohort.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proved NALD cohort:

  1. age 18 to 75 years
  2. receiving liver biopsy at the time of metabolic surgery
  3. relatively complete clinical information, including physical examination, biochemical and haematological assessments
* longitudinal cohort

  1. age 18 to 75 years
  2. receiving abdominal imaging examinations,
  3. relatively complete clinical information, including physical examination, biochemical and haematological assessments (4）follow-up time at least more than 12 months

Exclusion Criteria:

* (1)consumed excessive alcohol (≥140 g/week for males or ≥ 70 g/week for females) •
* (2) with history of other liver diseases including chronic hepatitis, biliary obstructive diseases or autoimmune hepatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study enrolled subjects who underwent liver biopsy or physical examination in Drum Tower Hospital affiliated to Nanjing University Medical School.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01-05 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Ischemic heart disease | up to 5 years
  Objective Findings of Coronary Stenosis (≥ 50%) in at least 2 coronary artery territories (ie, left anterior descending, ramus intermedius, left circumflex, right coronary artery) involving the vain vessel, a major branch, or a bypass graft
Documented heart disease checklist | up to 5 years
  Documented Myocardial Infarction or Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting
histological cirrhosis checklist | up to 5 years
  cirrhosis was defined as widespread disruption of normal liver structure by the formation of pseudolobules or Scheuer stage 4 fibrosis in pathological findings.
hepatocellular carcinoma | up to 5 years
  the diagnosis of hepatocellular carcinoma was based on well-established diagnostic imaging criteria and/or histology.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No